CLINICAL TRIAL: NCT04364243
Title: Pilot Study on Digitally Supported Home Exercises for the Management of Unspecific Low Back Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: ETH Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: BASEC-Nr: 2018-02132
Record Dates: First submitted 2019-10-30; First posted 2020-04-28 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: 2 x 2. Stratified randomization are used to assign patients to groups A and B and participants not receiving treatment to groups C and D. Participants are stratified by an average height.
Who Masked: Outcomes Assessor
Masking Description: Participants will be informed, instructed and provide consent to the study assistant, while assessments will be taken by a measurement assistant, blinded to the group assignment. Data which is not collected in all groups (e.g. intervention adherence) will be collected and managed by the study assistant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patients exercise (Experimental): Low back pain patients Next to basic medical physical training therapy group A receive a home exercising programme which involves 10 exercises for 2 minutes each with the Valedo training system.
  Interventions: Other: Digitally supported home exercises
- Patients control (No Intervention): Low back pain patients Group B will receive basic medical physical training therapy
- Non-patients exercise (Experimental): non-patients Groups C will receive a home exercising programme which involves 10 exercises for 2 minutes each with the Valedo training system.
  Interventions: Other: Digitally supported home exercises
- Non-patients control (No Intervention): non-patients Group D will receive no intervention

INTERVENTIONS:
Other: Digitally supported home exercises — The training will comprise of 9 sessions (3 weekly) Each of the training sessions will last 20 minutes. This will result in a cumulative total intervention exercise time of 180 minutes.
  Other Names: Valedo home
  Arms: Non-patients exercise; Patients exercise

SUMMARY:
The overall purpose of the study is to investigate effect of Digitally Supported Home Exercises (DSHE) in different groups for which digitally supported interventions could be beneficial. Balance is altered in individuals with low back pain and requires intervention Thus, the investigators will focus on the effect of DSHE to improve postural balance.

DETAILED DESCRIPTION:
The investigators want to investigate whether a digitally supported exercise program can improve the balance of people with non-specific lower back pain. During the exercise program, a computer game at home is controlled with the help of sensors attached to the body. Second aim is to record the daily activities of the participants and compare them with the back pain.

The 120 participants in this study will be divided into four groups (A, B, C and D). In groups A and B 20 patients are included who are in treatment for chronic back pain and receive Medical Training Therapy (MTT). For groups C and D the investigators will invite each 40 participants who have back pain but are not in treatment for their back pain. Only participants in groups A and C receive the digitally supported home exercise program. Who gets the training program is randomized using stratified block randomization.

The balance of all participants is measured four times. Between the 2nd and 3rd measurement the digitally supported exercise program is carried out. Between the 3rd and 4th assessement, participants in group A and C can exercise as much as they wish. The person who carries out the balance tests will not be informed which participant is in which group.

ELIGIBILITY:
Inclusion Criteria Group A and B

* Patients with chronic unspecific low back pain
* Patients of the Medical Training Therapy (MTT)
* Adult male and female participant's (≥18 years)
* Informed consent as documented by signature

Inclusion Criteria Group C and D

* Participant reports unspecific low back pain
* Receiving no therapy nor medical treatment for the last 6 months
* Adult male and female participant's (≥18 years)
* Informed consent as documented by signature

Exclusion criteria All Groups

* Patients with specific causes for low back pain
* Radicular syndrome
* Unable to participate currently in the program due to pain
* Pregnancy
* Medication effecting postural balance
* Uncorrected heavy visual impairment
* Allergy to adhesive tape
* Unable to understand and communicate in German or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
Postural Balance | At baseline (pretest 1), 3 weeks after pretest 1 (pretest 2), 3 weeks after pretest 2 (posttest 1), 6 weeks after posttest 1 (posttest2)
  Change of postural sway in anterior- posterior direction. Larger sway indicates worse balance. During each visit, 4 assessment repetitions of each 120 seconds are performed.

SECONDARY OUTCOMES:
Motor Control | At baseline (pretest 1), 3 weeks after pretest 1 (pretest 2), 3 weeks after pretest 2 (posttest 1), 6 weeks after posttest 1 (posttest 2)
  Lumbar spine and hip angles during task performance. Larger lumbar spine angles describe worse performance. Performance is assessed during a box lifting task and a waiter's bow task. At each assessment visit 5 repetitions of each task are performed.
Low back pain intensity | At balseline (pretest 1), 3 weeks after pretest 1 (pretest 2), 3 weeks after pretest 2 (posttest 1), 6 weeks after posttest 1 (posttest 2)
  Numeric rating scale (0-10), 0 = no pain, 10 = worst imaginable pain
Disability | At baseline (pretest 1), 3 weeks after pretest 1 (pretest 2), 3 weeks after pretest 2 (posttest 1), 6 weeks after posttest 1 ( posttest 2)
  The Roland-Morris Disability Questionnaire (RMDQ) is used to assess disability. Scores range from 0 to 24, with a value of 24 indicating higher disability
Health quality of life | At baseline (pretest 1), 3 weeks after pretest 1 (pretest 2), 3 weeks after pretest 2 (posttest 1), 6 weeks after posttest 1 (posttest 2)
  The short version of the World Health Organization Quality of Life Questionnaire (WOOQOL-BREF) is used to assess quality of Life. The scale has 4 subscales (raw scores range from 7 to 35, 6 to 30, 3 to 15 and 8 to 38). Larger values describe the better quality of life.
Fear of movement | At baseline (pretest 1), 3 weeks after pretest 1 (pretest 2), 3 weeks after pretest 2 (posttest 1), 6 weeks after posttest 1 (posttest 2)
  The short version of the Tampa Scale for Kinesiophobia (TSK-11) Questionnaire is used to assess fear of movement. The TSK-11 scores range from 11 to 44, with higher scores describing higher fear of movement.
Fear of specific movements | At baseline (pretest 1), 3 weeks after pretest 1 (pretest 2), 3 weeks after pretest 2 (posttest 1), 6 weeks after posttest 1 (posttest 2)
  Ratings of six movements (forward bending, backward bending, sideways bending, rotating, lifting a box, stretching upward) on each how painful or harmful a movement is and how careful a person is when executing the movement. Ratings range from 0 to 100. Large numbers indicate higher painfulness, fearfulness or caution when executing each movement.
Self-efficacy for managing chronic diseases | At baseline (pretest 1), 3 weeks after pretest 1 (pretest 2), 3 weeks after pretest 2 (posttest 1), 6 weeks after posttest 1 (posttest 2)
  Self-efficacy for managing chronic disease 6-item scale (SES-6) Questionnaire. The mean scores are interpreted and are between 1 and 10. Higher values are the better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jaap Swanenburg, PhD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Directorate of Research and Education, Physiotherapy & Occupational Therapy Research, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
Publication

REFERENCES:
- [Derived] Meinke A, Peters R, Knols RH, Swanenburg J, Karlen W. Feedback on Trunk Movements From an Electronic Game to Improve Postural Balance in People With Nonspecific Low Back Pain: Pilot Randomized Controlled Trial. JMIR Serious Games. 2022 Jun 10;10(2):e31685. doi: 10.2196/31685. PMID 35687390